CLINICAL TRIAL: NCT02009423
Title: A Prospective, Multicenter, Randomised, Double-blinded, Placebo-controlled, Two-parallel Groups, Phase III Study to Compare the Efficacy and Safety of Masitinib to Placebo in Patients With Localized, Primary Gastrointestinal Stromal Tumor (GIST) After Complete Surgery and With High Risk of Recurrence
Brief Title: Masitinib in Patients With Localized, Primary GIST After Complete Surgery and With High Risk of Recurrence
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision based on portfolio prioritization
Sponsor: AB Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AB12004
Record Dates: First submitted 2013-11-28; First posted 2013-12-12 (Estimated); Last update posted 2018-12-14 (Actual); Status verified 2018-12

CONDITIONS: Gastro-Intestinal Stromal Tumour
Keywords: Gastro-Intestinal Stromal Tumour; GIST; Localized primary tumor; Adjuvant therapy.
MeSH Terms: interventions — masitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Masitinib (Experimental): masitinib-treatment arm
  Interventions: Drug: Masitinib
- Placebo (Placebo Comparator): placebo-treatment arm
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Masitinib
  Arms: Masitinib
Drug: Placebo
  Arms: Placebo

SUMMARY:
The objective is to compare the efficacy and safety of masitinib at 4.5 mg/kg/day to placebo in the treatment of patients with localized, primary gastrointestinal stromal tumor (GIST) after complete surgery and with high risk of recurrence.

DETAILED DESCRIPTION:
Masitinib is a selective tyrosine kinase inhibitor with potent activity against wild-type c-Kit, the juxta membrane domain of c-Kit, and PDGFR. Masitinib is also thought to promote survival via modulation of immunostimulation-mediated anticancer effects and modulation of the tumor microenvironment. The objective is to compare the efficacy and safety of masitinib at 4.5 mg/kg/day with respect to placebo in the treatment of patients with localized, primary gastrointestinal stromal tumor (GIST) after complete surgery and with high risk of recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with histologic diagnosis of localized, primary GIST
2. Patient with measurable primary tumor lesion using conventional techniques or spiral CT scan assessed before tumor resection
3. Patient stopped imatinib as adjuvant therapy without progression OR patient not eligible for imatinib as adjuvant therapy
4. Patient with a high risk of recurrence, i.e., patients with primary tumor diameter > 5 cm and mitotic count > 5/50 HPF, or tumor diameter > 10 cm and any mitotic count, or tumor of any size with mitotic count > 10/50 HPF, or tumors that have ruptured into the peritoneal cavity
5. Patient without peritoneal or distant metastasis
6. Patient with c-kit (CD117) positive primary tumor detected immuno-histochemically
7. Patient after gross tumor resection (regardless of microscopic margins) within the past 14-70 days after surgery (R0 resection: negative microscopic margins or R1 resection: positive microscopic margins)
8. Patient free of tumor by post-operative imaging that included a baseline chest x-ray (or chest CT) and a post-operative abdomen and pelvis CT scan with intravenous and oral contrast or MRI with intravenous contrast within 28 days before the randomization
9. Patient with ECOG ≤ 2
10. Patient with adequate organ functions:

    * Absolute neutrophils count (ANC) ≥ 1.5 x 109/L
    * Hemoglobin ≥ 10 g/dL
    * Platelets (PTL) ≥ 75 x 109/L
    * AST/ALT ≤ 3x ULN
    * Gamma GT < 2.5 x ULN
    * Bilirubin ≤ 1.5x ULN
    * Normal creatinine or if abnormal creatinine, creatinine clearance ≥ 50 mL/min (Cockcroft and Gault formula)
    * Albumin > 1 x LLN
    * Proteinuria < 30 mg/mL (1+) on the dipstick. If proteinuria is ≥ 1+ on the dipstick, 24 hours proteinuria must be < 1.5g/24 hours
11. Patient with life expectancy > 3 months
12. Male or female patient, age >18 years
13. Patient weight > 40 kg and BMI > 18 kg/m²
14. Male and female patient of child bearing potential must agree to use two methods (one for the patient and one for the partner) of medically acceptable forms of contraception during the study and for 3 months after the last treatment intake. Female patient of child bearing potential must have a negative pregnancy test at screening and baseline
15. Patient able and willing to comply with study procedures as per protocol
16. Patient able to understand the patient card and to follow the patient card procedures in case of signs or symptoms of severe neutropenia or severe cutaneous toxicity, during the first 2 months of treatment
17. Patient able to understand, sign, and date the written informed consent form at the screening visit prior to any protocol-specific procedures are performed. If the patient is deemed by the treating physician to be cognitively impaired or questionably impaired in such a way that the ability of the patient to give informed consent is questionable, the designated legal guardian must sign the informed consent
18. Patient covered by insurance

Exclusion Criteria:

1. Patient with metastases of the primary GIST tumor
2. Patient treated for a cancer other than GIST within 5 years before enrolment, with the exception of basal cell carcinoma or cervical cancer in situ
3. Patient progressed under imatinib as adjuvant therapy
4. Patient with active central nervous system (CNS) metastasis or with history of CNS metastasis
5. Patient presenting with cardiac disorders defined by at least one of the following conditions:

   * Patient with recent cardiac history (within 6 months) of:

     * Acute coronary syndrome
     * Acute heart failure (class III or IV of the NYHA classification)
     * Significant ventricular arrhythmia (persistent ventricular tachycardia, ventricular fibrillation, resuscitated sudden death)
   * Patient with cardiac failure class III or IV of the NYHA classification
   * Patient with severe conduction disorders which are not prevented by permanent pacing (atrio-ventricular block 2 and 3, sino-atrial block)
   * Syncope without known etiology within 3 months
   * Uncontrolled hypertension or symptomatic hypertension, where hypertension is defined by systolic blood pressure > 140 mmHg or diastolic blood pressure > 90 mmHg and uncontrolled means that SBP lower than 140 mmHg and DBP lower than 90 mmHg are not achieved despite anti-hypertensive drugs, whatever the reason of failure (inadequate treatment, poor compliance, secondary hypertension or resistant hypertension).
6. Patient with history of poor compliance or history of drug/alcohol abuse, or excessive alcohol beverage consumption that would interfere with the ability to comply with the study protocol, or current or past psychiatric disease that might interfere with the ability to comply with the study protocol or give informed consent
7. Pregnant, or nursing female patient

Previous treatment

1. Patient previously treated with chemotherapy, radiation therapy, or investigational treatment following surgery

Wash-out

1. Treatment with any investigational agent within 4 weeks prior to Baseline visit
2. For patients treated with imatinib as adjuvant therapy, end of imatinib treatment must be between 5 days and 12 weeks prior to baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Recurrence Free Survival (RFS) | Until tumor recurrence (e.g. up to 24 months)
  e.g. from date of randomization until the date of first documented progression

SECONDARY OUTCOMES:
Overall Survival (OS) | until death of the patient (e.g. up to 24 months)
  e.g. from the date of randomization to the date of documented death